CLINICAL TRIAL: NCT05424354
Title: Prospective Randomized Open Label Multicenter Phase IV Clinical Trial to Compare Transforming Powder Dressing (TPD) to Current Standard of Care (SOC) Dressing Therapies in Acute Partial Thickness Burn Wounds
Brief Title: Acute Partial Thickness Burn Study Comparing Transforming Powder Dressing to Standard of Care Dressing
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ULURU Inc. (Industry)
Collaborators: Navy Advanced Medical Development (NAMD) Command (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-C-TPD-2021-02
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Wounds and Injuries
Keywords: burn
MeSH Terms: conditions — Wounds and Injuries; Burns

STUDY DESIGN:
Intervention Model Description: Randomized, Prospective, Multi-Center, Open Label, Comparison, Human, Interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transforming Powder Dressing (Experimental): Half of the subjects will be randomized to Transforming Powder Dressing (TPD) to treat the burn wound(s). Subjects will be evaluated on Treatment Day 0, 3, 7, 10, 14, 21, and 28 (or sooner if the wound heals prior to end of study visit on Day 28). On each study visit, wound care will be performed. TPD will be applied directly on the burn wound, followed by another dressing (often called a secondary dressing).
  Interventions: Device: Altrazeal (R) Transforming Powder Dressing
- Standard of Care Dressing (Active Comparator): Half of the subjects will be randomized to Standard of Care (SOC) to treat the burn wound(s). Subjects will be evaluated on Treatment Day 0, 3, 7, 10, 14, 21, and 28 (or sooner if the wound heals prior to end of study visit on Day 28). On each study visit, wound care will be performed. The standard of care burn dressing will be applied directly on the burn wound, followed by another dressing (often called a secondary dressing).
  Interventions: Other: Standard of Care burn dressing

INTERVENTIONS:
Device: Altrazeal (R) Transforming Powder Dressing — After informed consent and the subject is determined to meet all selection criteria, randomization will occur in a 1:1 ratio, to determine the treatment arm of the study. Half of those randomized will receive burn care with Altrazeal TPD.
  Arms: Transforming Powder Dressing
Other: Standard of Care burn dressing — After informed consent and the subject is determined to meet all selection criteria, randomization will occur in a 1:1 ratio, to determine the treatment arm of the study. Half of those randomized will receive burn care with the institution's standard of care burn dressing.
  Arms: Standard of Care Dressing

SUMMARY:
This study is being performed to assess the effectiveness of Altrazeal(R) Transforming Powder Dressing (TPD) in patients with partial thickness burns compared to the current standard of care (SOC) dressing. Adult men and women 18-65 years old who are hospitalized with an acute (meaning the burn injury occurred less than 72 hours prior to enrollment in the study) partial thickness burn wound, less than 20 percent of total body surface area may be considered. Subjects will be randomized in a 1:1 ratio to either SOC or TPD. Subjects will be followed for up to 28 days after enrollment.

DETAILED DESCRIPTION:
This post-marketing study is being performed to assess the effectiveness of Altrazeal(R) Transforming Powder Dressing (TPD) in patients with partial thickness burns compared to the current standard of care (SOC) dressing for burn wounds. Adult men and women 18-65 years old who are hospitalized with an acute (meaning the burn injury occurred less than 36 hours prior to enrollment in the study) partial thickness burn wound, comprising less than 20 percent of total body surface area may be considered. Subjects will be randomized in a 1:1 ratio to either SOC or TPD. Subjects will be followed during hospitalization and then upon discharge from the hospital for up to 28 days after enrollment into the study. At each of the 8 study visits, the burn wound will be evaluated, photographed and measured. The wound will be cleaned and debrided, if needed, per usual standard burn care. A wound dressing will be applied using TPD or a typical SOC dressing. Wound healing and wound pain will be monitored at each visit, and the results of the two groups (TPD and SOC) will be compared to each other. A survey evaluating the satisfaction with the dressing received will be given at the end of the study, or when the wound heals, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients who are receiving burn care; patients may be discharged when clinically stable and continue with outpatient treatment.
* Men and women (women cannot be pregnant or breast feeding) ages 18-65 years old
* Wounds must be partial thickness, involving up to 20% of the total body surface area.
* Burn injury should be less than 72 hours old
* Willing and able to comply with protocol mandated scheduled study visits/clinical evaluations.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Known allergy to TPD or its components

  * Women who are pregnant, breast feeding, or plan to get pregnant during the study period.
* Infected wounds
* Presence of any full thickness (third degree) burns
* Electrical burns
* Heavily draining burns due to underlying chronic lymphedema or other conditions
* Concurrent clinical condition within the judgement of the clinician, pose a health risk to the patient, delay wound healing, or otherwise influence the outcome of the study.
* History of poor wound healing and/or skin/immune system condition

  * Deemed by clinician not to be suitable
* Unwilling or not able to provide consent or comply with protocol or required visits
* Developmental disability/significant psychological disorder which can impair the subjects ability to provide informed consent, or participate in the study protocol
* Active alcohol or substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain from the Burn Wound | 28 days (or sooner if the wound heals prior to 28 days)
  Subjects will complete a visual analogue scale (VAS) to rate their pain prior to, during and after dressing changes. The scale ranges from 0 to 10, with 0 indicating no pain and 10 indicating the worst pain possible.

SECONDARY OUTCOMES:
Wound healing | 28 days (or sooner if the wound heals prior to 28 days)
  Wounds will measured at each study visit to determine surface area healing.
Safety of the Interventions (TPD and SOC) | 28 days (or sooner if the wound heals prior to 28 days)
  Complications such as infection, and other adverse events that develop will be documented, evaluated for severity, and compared between intervention groups.
Subject satisfaction | End of Study
  Subjects will be asked to complete a subject satisfaction survey, which consists of 8 multiple choice questions regarding their wound dressing.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Saxe, MD, Principal Investigator — ULURU Inc.
Locations (6):
- United States (6):
  - University of California-Irvine, Orange, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Jackson Memorial Hospital UM/JMH Burn Center, Miami, Florida
  - University of Louisville Health, Louisville, Kentucky
  - Westchester Medical Center, Valhalla, New York
  - University of Texas SW (Parkland), Dallas, Texas

IPD SHARING:
Plan to Share IPD: No